CLINICAL TRIAL: NCT05531799
Title: Optimizing an Anal High-grade Squamous Intraepithelial Lesion Screening Algorithm for Thai Men Who Have Sex With Men and Transgender Women
Brief Title: Anal HSIL Screening Algorithm
Acronym: 0007/65
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of HIV Research and Innovation Foundation, Thailand (Other)
Collaborators: National Institutes of Health (NIH) (NIH); amfAR, The Foundation for AIDS Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Screening
Other Study IDs: IHRI013
Record Dates: First submitted 2022-06-08; First posted 2022-09-08 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Anal High-grade Squamous Intraepithelial Lesion
Keywords: Anal cytology; Human papillomavirus(HPV); High resolution anoscopy (HRA)

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (12):
- Group 1 DARE/CYTOLOGY/HPV/HRA (Other): Participant request physician assessment for Digital anal rectal exam, Anal cytology, Anal HPV test and High resolution anoscopy for every 6 months within 12 months period
  Interventions: Procedure: OPTIMIZATION PHASE
- Group 2 DARE/CYTOLOGY/HPV (Other): Participant request physician assessment for Digital anal rectal exam, Anal cytology, Anal HPV test for every 6 months within 12 months period
  Interventions: Procedure: OPTIMIZATION PHASE
- Group 3 DARE/CYTOLOGY/HRA (Other): Participant request physician assessment for Digital anal rectal exam, Anal cytology and High resolution anoscopy for every 6 months within 12 months period
  Interventions: Procedure: OPTIMIZATION PHASE
- Group 4 DARE/CYTOLOGY (Other): Participant request physician assessment for Digital anal rectal exam, Anal cytology for every 6 months within 12 months period
  Interventions: Procedure: OPTIMIZATION PHASE
- Group 5 DARE/HPV/HRA (Other): Participant request physician assessment for Digital anal rectal exam, Anal HPV test and High resolution anoscopy for every 6 months within 12 months period
  Interventions: Procedure: OPTIMIZATION PHASE
- Group 6 DARE/HPV (Other): Participant request physician assessment for Digital anal rectal exam and Anal HPV test for every 6 months within 12 months period
  Interventions: Procedure: OPTIMIZATION PHASE
- Group 7 DARE/HRA (Other): Participant request physician assessment for Digital anal rectal exam and High resolution anoscopy for every 6 months within 12 months period
  Interventions: Procedure: OPTIMIZATION PHASE
- Group 8 DARE (Other): Participant request physician assessment for Digital anal rectal exam for every 6 months within 12 months period
  Interventions: Procedure: OPTIMIZATION PHASE
- Self-collection CYTOLOGY/HPV (Other): Participant request Self-sampling collection for Anal cytology and Anal HPV test for every 6 months within 12 months period
  Interventions: Procedure: OPTIMIZATION PHASE
- Self-collection CYTOLOGY (Other): Participant request Self-sampling collection for Anal cytology for every 6 months within 12 months period
  Interventions: Procedure: OPTIMIZATION PHASE
- Self-collection HPV (Other): Participant request Self-sampling collection for Anal HPV test for every 6 months within 12 months period
  Interventions: Procedure: OPTIMIZATION PHASE
- Self-collection control group CYTOLOGY/HPV (Other): Participant request Self-sampling collection for Anal cytology and Anal HPV only at month 12
  Interventions: Procedure: OPTIMIZATION PHASE

INTERVENTIONS:
Procedure: OPTIMIZATION PHASE — The goal of the optimization phase of MOST is to identify the most promising combination of experimental components in changing an outcome given a set of environmental constraints. Looking at effectiveness, efficiency, economy, and scalability criteria, we will focus on the proportion of anal HSIL identified (effectiveness), unit cost (efficiency and economy), and accumulating cost to the client over a 12-month period (economy). Meeting these criteria will likely imply scalability. The most appropriate anal HSIL screening algorithm would ideally be one which could
  - identify anal HSIL in at least 20% of HIV-positive MSM and 10% of HIV-negative MSM at baseline and

SUMMARY:
This the propose to use the Multiphase Optimization Strategy Trial (MOST) design to identify an anal HSIL screening algorithm which is most suitable in terms of effectiveness, efficiency, and economy. Specifically, The Investigators will use a factorial design as the main strategy in the MOST, as this allows the evaluation of multiple intervention components that are candidates for ultimate inclusion in the algorithm. The Investigators will then implement the most suitable anal HSIL screening algorithm in the clinic, using the RE-AIM (Reach, Effectiveness, Adoption, Implementation, Maintenance) framework to guide its design, implementation, and evaluation. An interrupted time series will be used to compare anal HSIL screening uptake among men who have sex with men clients in the clinic, prior to and after the implementation of the new anal HSIL screening algorithm, and mixed-methods approaches will be used to evaluate components of the RE-AIM framework.

DETAILED DESCRIPTION:
I. PREPARATION PHASE Purpose To lay groundwork for optimization of anal high-grade squamous intraepithelial lesion screening algorithm for MSM, and identify which test and component(s) should be included in the anal HSIL screening algorithm.

II. OPTIMIZATION PHASE Purpose To form an anal high-grade squamous intraepithelial lesion screening algorithm that meets the optimization criteria.

III. EVALUATION PHASE Purpose To establish whether the optimized anal high-grade squamous intraepithelial lesion screening algorithm has a statistically significant effect on service uptake among MSM compared to the standard of care.

ELIGIBILITY:
Inclusion criteria

Clients for MSM and TGW:

* Thai nationality, men with self-identifies as MSM and/or TGW
* HIV-positive MSM/TGW aged 30 years or older or
* HIV-negative MSM/TGW aged 40 years or older

Clinic staff:

- Has worked in the study clinic during phase III

Government stakeholders:

- Involved in health policy development in Thailand

Exclusion criteria

Clients for MSM and TGW:

* Unable to perform any study procedures, or unable to commit to attend all study visits.
* Had Anal cancer lesion at enrollment visit, this exclusion for participation in phase II study.

Clinic staff:

- Not willing to participate in the evaluation

Government stakeholders:

- Not willing to participate in the evaluation

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 950 (Estimated)
Dates: Start 2022-05-18 (Actual); Primary Completion 2027-12-20 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
Identify new cases of anal HSIL by Anal HSIL screening algorithm | 18 months
  identify anal HSIL in at least 20% of HIV-positive MSM/TGW and 10% of HIV-negative MSM/TGW within visit schedule.
Compare anal HSIL screening method to new anal HSIL screening method algorithm | 24 months
  Evaluate anal HSIL screening method uptake among MSM/TGW clients in the clinic compare to the implementation of the new anal HSIL screening method algorithm.

CONTACTS AND LOCATIONS:
Overall Officials: Nittaya Phanuphak, MD,PhD., Principal Investigator — Institute of HIV Research and Innovation
Locations (1):
- Institute of HIV Research and Innovation, Pathum Wan, Bangkok, Thailand